CLINICAL TRIAL: NCT05375994
Title: A Phase 1/2 Study of Avutometinib (VS-6766) in Combination With Adagrasib in Patients With KRAS G12C Mutant Non-Small Cell Lung Cancer (NSCLC) (RAMP 204)
Brief Title: Study of Avutometinib (VS-6766) + Adagrasib in KRAS G12C NSCLC Patients
Acronym: RAMP204
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Collaborators: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VS-6766-204
Record Dates: First submitted 2022-05-02; First posted 2022-05-17 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Non Small Cell Lung Cancer; KRAS Activating Mutation; Advanced Cancer; Metastatic Cancer; Malignant Neoplasm of Lung; Malignant Neoplastic Disease
Keywords: NSCLC; KRAS G12C; Non Small Cell Lung Cancer; Metastatic Cancer; Adagrasib; Avutometinib (VS-6766)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms; Neoplasms | interventions — adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- avutometinib(VS-6766)+adagrasib (Experimental): To determine the recommended phase 2 dose (RP2D) for VS-6766 in combination with adagrasib in G12C inhibitor exposed patients
  Interventions: Drug: avutometinib (VS-6766) and adagrasib
- avutometinib (VS-6766)+adagrasib RP2D (Experimental): To determine the efficacy of the RP2D identified from Part A in G12C inhibitor exposed patients
  Interventions: Drug: avutometinib (VS-6766) and adagrasib

INTERVENTIONS:
Drug: avutometinib (VS-6766) and adagrasib — The RP2D of VS-6766 + adagrasib determined in Part A will be used in Part B dose expansion
  Other Names: KRAS G12C Inhibitor, adagrasib, KRAZATI®

SUMMARY:
This study will assess the safety and efficacy of avutometinib (VS-6766) in combination with adagrasib in patients with G12C Non-Small Cell Lung Cancer (NSCLC) who have been exposed to prior G12C inhibitor and experienced progressive disease.

DETAILED DESCRIPTION:
This is a multicenter, non-randomized, open-label Phase 1/2 study designed to evaluate safety, tolerability and efficacy of avutometinib (VS-6766) in combination with adagrasib in patients with KRAS G12C mutant NSCLC who have been exposed to prior G12C inhibitor and experienced progressive disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years of age
* Histologic or cytologic evidence of NSCLC
* Known KRAS G12C mutation
* The subject must have received prior therapy with a KRAS G12C inhibitor and experienced progression
* Must have received appropriate treatment with at least one prior systemic regimen, but no more than 3 prior regimens, for Stage 3B-C or 4 NSCLC
* Measurable disease according to RECIST 1.1
* An Eastern Cooperative Group (ECOG) performance status ≤ 1
* Adequate organ function
* Adequate recovery from toxicities related to prior treatments
* Agreement to use highly effective method of contraceptive

Exclusion Criteria:

* Prior chemotherapy, targeted therapies, radiotherapy, immunotherapy or treatment with an investigational agent within 14 days of receipt of study drug (within 6 weeks for nitrosoureas, mitomycin C and chest radiation; within 6 months prior to Cycle 1 Day 1 for chest radiation > 30Gy)
* History of prior malignancy, with the exception of curatively treated malignancies
* Major surgery within 4 weeks (excluding placement of vascular access)
* Exposure to strong CYP3A4 inhibitors or inducers within 14 days prior to the first dose and during the course of therapy
* Exposure to strong inhibitors of breast cancer resistance protein (BCRP) within 14 days prior to the first dose and during the course of therapy
* Symptomatic brain metastases requiring steroids or other local interventions within the 2 weeks prior to initiation of therapy
* Known SARS-Cov2 infection ≤28 days prior to first dose of study therapy
* Known hepatitis B, hepatitis C, or human immunodeficiency virus infection that is active
* Active skin disorder that has required systemic therapy within the past 1 year
* History of rhabdomyolysis or interstitial lung disease
* Concurrent ocular disorders
* Concurrent heart disease or severe obstructive pulmonary disease
* Subjects with the inability to swallow oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Part A: To determine RP2D for avutometinib(VS-6766) in combination with adagrasib | From start of treatment to confirmation of RP2D; 28 days
  Assessment of Dose-limiting toxicities (DLTs)
To determine the efficacy of the optimal regimen identified from Part A | From start of treatment to confirmation of response; 16 weeks
  Confirmed overall response rate per RECIST 1.1

SECONDARY OUTCOMES:
To characterize the safety and toxicity profile: | 24 Months
  * Incidence of Adverse events (AEs) and Serious Adverse Events (SAEs) assessed by the toxicity grading of the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v 5.0)
  * Severity of Adverse events (AEs) and Serious Adverse Events (SAEs) by toxicity grade assessed by the toxicity grading of the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v 5.0)
  * Duration of Adverse events (AEs) and Serious Adverse Events (SAEs)
  * Incidence of clinically significant changes in lab parameters
  * Incidence of abnormal vital signs (including systolic and diastolic blood pressure in mmHg)
ECG QT Interval | 24 months
  Corrected ECG QT interval by Fredericia (QTcF)
Duration of Response (DOR) | Time from the first documentation of response to first documentation of progressive disease or death due to any cause, greater than or equal to 6 months
  Time of first response to PD as assessed per RECIST 1.1
Disease Control Rate (DCR) | Greater than or equal to 8 weeks
  CR and PR stable disease as assessed per RECIST 1.1
Progression Free Survival (PFS) | 24 months
  From the time of first dose of study intervention to PD or death from any cause
Overall Survival (OS) | Up to 5 years
  From time of first dose of study intervention to death
Plasma Pharmacokinetics (PK) of avutometinib(VS 6766), adagrasib, and relevant metabolites - Tmax | 10 weeks
  time of Maximum concentration (Tmax)
Plasma Pharmacokinetics (PK) of avutometinib(VS 6766), adagrasib, and relevant metabolites - AUC | 10 weeks
  Area under plasma Concentration (AUC) 0 to t
Plasma Pharmacokinetics (PK) of avutometinib(VS 6766), adagrasib, and relevant metabolites - Half-life | 10 weeks
  concentration Half-life (T1/2)
Clinical Benefit Rate | ≥ 6 months
  defined as Complete Response+Partial Response +Stable Disease

CONTACTS AND LOCATIONS:
Overall Officials: MD Verastem, Study Director — Verastem, Inc.
Locations (8):
- United States (8):
  - UCSF Thoracic Oncology, San Francisco, California
  - University of Colorado Hospital Anschutz Cancer Pavllion, Aurora, Colorado
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Virginia Cancer Specialists, NEXT Oncology, Fairfax, Virginia
  - Medical College Wisconsin, Milwaukee, Wisconsin